CLINICAL TRIAL: NCT05179785
Title: Establishing the Effect of Electroencephalography (EEG)-Guided Theta Burst Stimulation on Reducing Mania/Hypomania-related Affect and Reward Driven Behavior in Bipolar Disorder
Brief Title: Examining the Effect of EEG-guided Theta Burst Stimulation in Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mary Phillips, MD MD (Cantab) (Other)
Collaborators: Milken Institute (Other)
Responsible Party: Sponsor-Investigator, Mary Phillips, MD MD (Cantab), Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STUDY21110077
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Transcranial Magnetic Stimulation; Electroencephalography
MeSH Terms: conditions — Bipolar Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Left vLPFC cTBS/right dlPFC iTBS/left Som cTBS (Experimental): A random number sequence will be generated for randomization of the 3 EEG/TBS session order to which each participant is assigned:
  left vlPFC cTBS (cTBS applied to the left ventrolateral prefrontal cortex) right dlPFC iTBS (iTBS applied to the right dorsolateral prefrontal cortex) left Som cTBS (cTBS applied to the left somatosensory cortex)
  Interventions: Device: Continuous Theta Burst Stimulation (cTBS); Device: Intermittent Theta Burst Stimulation (iTBS)
- Left vLPFC cTBS/left Som cTBS/right dlPFC iTBS (Experimental): A random number sequence will be generated for randomization of the 3 EEG/TBS session order to which each participant is assigned:
  left vlPFC cTBS (cTBS applied to the left ventrolateral prefrontal cortex) left Som cTBS (cTBS applied to the left somatosensory cortex) right dlPFC iTBS (iTBS applied to the right dorsolateral prefrontal cortex)
  Interventions: Device: Continuous Theta Burst Stimulation (cTBS); Device: Intermittent Theta Burst Stimulation (iTBS)
- left Som cTBS/right dlPFC iTBS/Left vLPFC cTBS (Experimental): A random number sequence will be generated for randomization of the 3 EEG/TBS session order to which each participant is assigned:
  left Som cTBS (cTBS applied to the left somatosensory cortex) right dlPFC iTBS (iTBS applied to the right dorsolateral prefrontal cortex) left vlPFC cTBS (cTBS applied to the left ventrolateral prefrontal cortex)
  Interventions: Device: Continuous Theta Burst Stimulation (cTBS); Device: Intermittent Theta Burst Stimulation (iTBS)
- left Som cTBS/Left vLPFC cTBS/right dlPFC iTBS (Experimental): A random number sequence will be generated for randomization of the 3 EEG/TBS session order to which each participant is assigned:
  left Som cTBS (cTBS applied to the left somatosensory cortex) left vlPFC cTBS (cTBS applied to the left ventrolateral prefrontal cortex) right dlPFC iTBS (iTBS applied to the right dorsolateral prefrontal cortex)
  Interventions: Device: Continuous Theta Burst Stimulation (cTBS); Device: Intermittent Theta Burst Stimulation (iTBS)
- right dlPFC iTBS/left Som cTBS/Left vLPFC cTBS (Experimental): A random number sequence will be generated for randomization of the 3 EEG/TBS session order to which each participant is assigned:
  right dlPFC iTBS (iTBS applied to the right dorsolateral prefrontal cortex) left Som cTBS (cTBS applied to the left somatosensory cortex) left vlPFC cTBS (cTBS applied to the left ventrolateral prefrontal cortex)
  Interventions: Device: Continuous Theta Burst Stimulation (cTBS); Device: Intermittent Theta Burst Stimulation (iTBS)
- right dlPFC iTBS/Left vLPFC cTBS/left Som cTBS (Experimental): A random number sequence will be generated for randomization of the 3 EEG/TBS session order to which each participant is assigned:
  right dlPFC iTBS (iTBS applied to the right dorsolateral prefrontal cortex) left vlPFC cTBS (cTBS applied to the left ventrolateral prefrontal cortex) left Som cTBS (cTBS applied to the left somatosensory cortex)
  Interventions: Device: Continuous Theta Burst Stimulation (cTBS); Device: Intermittent Theta Burst Stimulation (iTBS)

INTERVENTIONS:
Device: Continuous Theta Burst Stimulation (cTBS) — cTBS is a brief stimulation of a part of the brain with a magnetic field that passes through the scalp and skull safely that can decrease the excitability of cortical neurons. It is FDA-approved as a treatment for psychological conditions including depression; however, this device is not approved for the treatment of adults with Bipolar Disorder I or for use in healthy adults. This research study is using the cTBS off label in all participants (those with and without Bipolar Disorder I) to examine research questions
  Other Names: Transcranial Magnetic Stimulation (TMS)
Device: Intermittent Theta Burst Stimulation (iTBS) — iTBS is a brief stimulation of a part of the brain with a magnetic field that passes through the scalp and skull safely to increase the excitability of cortical neurons. It is FDA-approved as a treatment for psychological conditions including depression; however, this device is not approved for the treatment of adults with Bipolar Disorder I or for use in healthy adults. This research study is using the cTBS off label in all participants (those with and without Bipolar Disorder I) to examine research questions.
  Other Names: Transcranial Magnetic Stimulation (TMS)

SUMMARY:
Bipolar Disorder (BD) is a common and highly debilitating psychiatric disorder, however, the predisposing brain mechanisms are poorly understood. Here, the investigators will conduct a proof of concept study that will examine the effect of electroencephalography (EEG)-guided theta burst stimulation (TBS) on reducing mania/hypomania-related affect and reward driven behavior in adults with BD. The investigators hypothesize that TBS will reduce mania/hypomania-related affect and reward driven behavior in adults with BD.

DETAILED DESCRIPTION:
This study aims to examine the effect of electroencephalography (EEG)-guided theta burst stimulation (TBS) on reducing mania/hypomania-related affect and reward driven behavior in adults with BD. Eligible participants will undergo 6 study visits: a screening visit, a baseline MRI visit, TBS motor thresholding visit, and 3 cTBS/EEG visits. Participants will receive brain stimulation and have brain activity recorded by EEG at each of the 3 cTBS/EEG study visits. The research associates (except for the research associate administering the TBS) and participants will be blinded to the brain area receiving TBS, which will be randomized and counterbalanced beforehand. Certain information is withheld to protect the scientific integrity of the study design.

The goal of the study is to reduce overactivity in the reward neural network (RNet) and increase activity in the central executive control network (CEN) using theta burst stimulation (TBS). The region in the RNet to be targeted by inhibitory (continuous, cTBS) is the left ventrolateral prefrontal cortex (vlPFC); and the region in the CEN to be targeted by excitatory (intermittent, iTBS) is the right dorsolateral prefrontal cortex (dlPFC)

ELIGIBILITY:
Inclusion criteria:

* 18-35 years of age
* Diagnosis of BD (DSM-5 criteria) in remission (euthymic for >2 months) or in a manic/hypomanic episode [manic/hypomanic or euthymic adults with BD (3-fifths manic/hypomanic); euthymic for > 2 months from most recent BD episode OR current manic/hypomanic episode]
* Not psychotic
* Score <3 on delusions, hallucinations, unusual thought content, and conceptual disorganization items of the Positive and Negative Syndrome Scale (PANSS)
* Unmedicated or on any combination of anxiolytics (benzodiazepines, buspirone, pregabalin, hydroxyzine) as needed, and/or atypical antipsychotics, and/or lithium, and/or other mood stabilizers, and/or non-SNRI antidepressants and/or non benzodiazepine hypnotics, as these are commonly-prescribed medications for BD
* Provides the contact information of a medical provider (including but not limited to a PCP) that we may communicate with for any concerns of escalating symptoms of mania

Exclusion criteria:

* Not 18-35 years of age
* Diagnosis of BD in a depressive episode or Diagnosis of BP in partial remission, euthymia that fails to meet full remission criterion of a period of at least 2 months in which there are no significant symptoms, e.g., only partial remission of symptoms or full remission of symptoms but for <2 months
* Diagnosis of BD in a depressive episode
* Personal and family history of epilepsy (TBS exclusion)
* Binge alcohol drinking
* Taking substances in the last month that can elevate seizure risk including but not limited to SNRI antidepressants, bupropion and stimulants (TBS exclusion)
* History of head injury, neurological, pervasive developmental disorder (e.g. autism), systemic medical disease and treatment (medical records, participant report)
* Mini-Mental State Examination score (cognitive state) <24
* Premorbid NAART IQ estimate<85
* Visual disturbance: <20/40 Snellen visual acuity
* History of alcohol/substance use disorder (SUD; all substances, except nicotine), and/or illicit substance use (except cannabis) over the last 6 months (SCID-5). Note: lifetime/present cannabis use (at non-abuse (<3 times in the past month) and non SUD levels) will be allowed, given its common usage in BD and young adults. Cannabis SUD over the last 6 months will not be allowed. Urine tests on scan days will exclude current illicit substance use (except cannabis). Salivary alcohol tests on scan days will exclude intoxicated individuals
* Binge drinking in the week before, and/or >3 units/day for the 3 days before, and/or alcohol in the last 12 hrs before, any TBS visit, confirmed at screening and scan days (to avoid TBS during alcohol withdrawal). Alcohol/nicotine/ caffeine/cannabis use (below SCID-5 SUD, binge levels) will be allowed, and used as covariates
* MRI exclusion: metallic objects, e.g., surgical implants; claustrophobia; positive pregnancy test for females (at the MRRC) or self-report pregnancy *Unable to understand English
* Scoring greater than or equal to 8 on HRSD at screen visit and depressive episode is confirmed on SCID-5
* Scoring greater than or equal to 18 on HRSD at any study visit
* Psychosis
* Using psychotropic medications other than those allowed in inclusion criteria
* Scoring greater than or equal to 38 on the YMRS at any study visit
* Does not provide the contact information of a medical provider (including but not limited to a PCP) that we may communicate with for any concerns of escalating symptoms of mania

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary L Phillips, MD, MD, Principal Investigator — University of Pittsburgh; Fabio Ferrarelli, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Informed consent will be collected from study participants that allows for broad sharing of participants' de-identified data. Data transfer procedures will be in accordance with all Institutional Review Board guidelines and federal regulations including HIPAA.
Time Frame: The PIs reserve the right to publish on the stated aims in a timely manner during the period of the award. Data will be available for addressing other research questions (i.e. which are not described in funded/pending grants) as soon as the data have been checked for accuracy (a period which will be no later than one year after the completion of each assessment). After the award has ended, the study investigators will continue to test the stated aims, but will also continue to solicit collaborations with outside researchers and to consider data requests in a timely manner.
Access Criteria: Outside investigators must submit a 1)proposal of the study aims, hypotheses, variables/constructs, analytic approach, and estimated duration of the proposed research; 2)resume, qualifications, source of financial support, and conflict of interest statement; 3)sign a data-sharing agreement and confidentiality statement that stipulates using the data for the stated research purposes only, securing the data using appropriate computer technology, not manipulating the data in order to identify participants, acknowledging the grant that supported data collection and management in publications/presentations, and destroying or returning the data after analyses are complete; 4)obtain approval from their Institutional Review Board, and along with other staff members who have access to the data, submit certificates of the University of Pittsburgh Education and Certification Program in Research Practice Fundamentals or provide written documentation pf similar human subjects protection training.

REFERENCES:
- [Result] Mayeli A, Wang Y, Graur S, Ghane M, Keihani A, Kim A, Janssen S, Huston C, Coffman BA, Ferrarelli F, Phillips ML. Effects of theta burst stimulation on reward processing and decision-making in bipolar disorder: A pilot study. Brain Stimul. 2024 Mar-Apr;17(2):163-165. doi: 10.1016/j.brs.2024.02.002. Epub 2024 Feb 7. No abstract available. PMID 38336341

RESULTS

PARTICIPANT FLOW:
Groups:
- Left vLPFC cTBS/Right dlPFC iTBS/Left Som cTBS: A random number sequence will be generated for randomization of the 3 EEG/TBS session order to which each participant is assigned:
  left vlPFC cTBS (cTBS applied to the left ventrolateral prefrontal cortex) right dlPFC iTBS (iTBS applied to the right dorsolateral prefrontal cortex) left Som cTBS (cTBS applied to the left somatosensory cortex)
  Continuous Theta Burst Stimulation (cTBS): cTBS is a brief stimulation of a part of the brain with a magnetic field that passes through the scalp and skull safely that can decrease the excitability of cortical neurons. It is FDA-approved as a treatment for psychological conditions including depression; however, this device is not approved for the treatment of adults with Bipolar Disorder I or for use in healthy adults. This research study is using the cTBS off label in all participants (those with and without Bipolar Disorder I) to examine research questions
  Intermittent Theta Burst Stimulation (iTBS): iTBS is a brief stimulation of a part of the brain with a magnetic field that passes through the scalp and skull safely to increase the excitability of cortical neurons. It is FDA-approved as a treatment for psychological conditions including depression; however, this device is not approved for the treatment of adults with Bipolar Disorder I or for use in healthy adults. This research study is using the cTBS off label in all participants (those with and without Bipolar Disorder I) to examine research questions.
- Left vLPFC cTBS/Left Som cTBS/Right dlPFC iTBS: A random number sequence will be generated for randomization of the 3 EEG/TBS session order to which each participant is assigned:
  left vlPFC cTBS (cTBS applied to the left ventrolateral prefrontal cortex) left Som cTBS (cTBS applied to the left somatosensory cortex) right dlPFC iTBS (iTBS applied to the right dorsolateral prefrontal cortex)
  Continuous Theta Burst Stimulation (cTBS): cTBS is a brief stimulation of a part of the brain with a magnetic field that passes through the scalp and skull safely that can decrease the excitability of cortical neurons. It is FDA-approved as a treatment for psychological conditions including depression; however, this device is not approved for the treatment of adults with Bipolar Disorder I or for use in healthy adults. This research study is using the cTBS off label in all participants (those with and without Bipolar Disorder I) to examine research questions
  Intermittent Theta Burst Stimulation (iTBS): iTBS is a brief stimulation of a part of the brain with a magnetic field that passes through the scalp and skull safely to increase the excitability of cortical neurons. It is FDA-approved as a treatment for psychological conditions including depression; however, this device is not approved for the treatment of adults with Bipolar Disorder I or for use in healthy adults. This research study is using the cTBS off label in all participants (those with and without Bipolar Disorder I) to examine research questions.
- Left Som cTBS/Right dlPFC iTBS/Left vLPFC cTBS: A random number sequence will be generated for randomization of the 3 EEG/TBS session order to which each participant is assigned:
  left Som cTBS (cTBS applied to the left somatosensory cortex) right dlPFC iTBS (iTBS applied to the right dorsolateral prefrontal cortex) left vlPFC cTBS (cTBS applied to the left ventrolateral prefrontal cortex)
  Continuous Theta Burst Stimulation (cTBS): cTBS is a brief stimulation of a part of the brain with a magnetic field that passes through the scalp and skull safely that can decrease the excitability of cortical neurons. It is FDA-approved as a treatment for psychological conditions including depression; however, this device is not approved for the treatment of adults with Bipolar Disorder I or for use in healthy adults. This research study is using the cTBS off label in all participants (those with and without Bipolar Disorder I) to examine research questions
  Intermittent Theta Burst Stimulation (iTBS): iTBS is a brief stimulation of a part of the brain with a magnetic field that passes through the scalp and skull safely to increase the excitability of cortical neurons. It is FDA-approved as a treatment for psychological conditions including depression; however, this device is not approved for the treatment of adults with Bipolar Disorder I or for use in healthy adults. This research study is using the cTBS off label in all participants (those with and without Bipolar Disorder I) to examine research questions.
- Left Som cTBS/Left vLPFC cTBS/Right dlPFC iTBS: A random number sequence will be generated for randomization of the 3 EEG/TBS session order to which each participant is assigned:
  left Som cTBS (cTBS applied to the left somatosensory cortex) left vlPFC cTBS (cTBS applied to the left ventrolateral prefrontal cortex) right dlPFC iTBS (iTBS applied to the right dorsolateral prefrontal cortex)
  Continuous Theta Burst Stimulation (cTBS): cTBS is a brief stimulation of a part of the brain with a magnetic field that passes through the scalp and skull safely that can decrease the excitability of cortical neurons. It is FDA-approved as a treatment for psychological conditions including depression; however, this device is not approved for the treatment of adults with Bipolar Disorder I or for use in healthy adults. This research study is using the cTBS off label in all participants (those with and without Bipolar Disorder I) to examine research questions
  Intermittent Theta Burst Stimulation (iTBS): iTBS is a brief stimulation of a part of the brain with a magnetic field that passes through the scalp and skull safely to increase the excitability of cortical neurons. It is FDA-approved as a treatment for psychological conditions including depression; however, this device is not approved for the treatment of adults with Bipolar Disorder I or for use in healthy adults. This research study is using the cTBS off label in all participants (those with and without Bipolar Disorder I) to examine research questions.
- Right dlPFC iTBS/Left Som cTBS/Left vLPFC cTBS: A random number sequence will be generated for randomization of the 3 EEG/TBS session order to which each participant is assigned:
  right dlPFC iTBS (iTBS applied to the right dorsolateral prefrontal cortex) left Som cTBS (cTBS applied to the left somatosensory cortex) left vlPFC cTBS (cTBS applied to the left ventrolateral prefrontal cortex)
  Continuous Theta Burst Stimulation (cTBS): cTBS is a brief stimulation of a part of the brain with a magnetic field that passes through the scalp and skull safely that can decrease the excitability of cortical neurons. It is FDA-approved as a treatment for psychological conditions including depression; however, this device is not approved for the treatment of adults with Bipolar Disorder I or for use in healthy adults. This research study is using the cTBS off label in all participants (those with and without Bipolar Disorder I) to examine research questions
  Intermittent Theta Burst Stimulation (iTBS): iTBS is a brief stimulation of a part of the brain with a magnetic field that passes through the scalp and skull safely to increase the excitability of cortical neurons. It is FDA-approved as a treatment for psychological conditions including depression; however, this device is not approved for the treatment of adults with Bipolar Disorder I or for use in healthy adults. This research study is using the cTBS off label in all participants (those with and without Bipolar Disorder I) to examine research questions.
- Right dlPFC iTBS/Left vLPFC cTBS/Left Som cTBS: A random number sequence will be generated for randomization of the 3 EEG/TBS session order to which each participant is assigned:
  right dlPFC iTBS (iTBS applied to the right dorsolateral prefrontal cortex) left vlPFC cTBS (cTBS applied to the left ventrolateral prefrontal cortex) left Som cTBS (cTBS applied to the left somatosensory cortex)
  Continuous Theta Burst Stimulation (cTBS): cTBS is a brief stimulation of a part of the brain with a magnetic field that passes through the scalp and skull safely that can decrease the excitability of cortical neurons. It is FDA-approved as a treatment for psychological conditions including depression; however, this device is not approved for the treatment of adults with Bipolar Disorder I or for use in healthy adults. This research study is using the cTBS off label in all participants (those with and without Bipolar Disorder I) to examine research questions
  Intermittent Theta Burst Stimulation (iTBS): iTBS is a brief stimulation of a part of the brain with a magnetic field that passes through the scalp and skull safely to increase the excitability of cortical neurons. It is FDA-approved as a treatment for psychological conditions including depression; however, this device is not approved for the treatment of adults with Bipolar Disorder I or for use in healthy adults. This research study is using the cTBS off label in all participants (those with and without Bipolar Disorder I) to examine research questions.
Period: Overall Study
Arm/Group | Left vLPFC cTBS/Right dlPFC iTBS/Left Som cTBS | Left vLPFC cTBS/Left Som cTBS/Right dlPFC iTBS | Left Som cTBS/Right dlPFC iTBS/Left vLPFC cTBS | Left Som cTBS/Left vLPFC cTBS/Right dlPFC iTBS | Right dlPFC iTBS/Left Som cTBS/Left vLPFC cTBS | Right dlPFC iTBS/Left vLPFC cTBS/Left Som cTBS
Started | 3 | 2 | 1 | 2 | 3 | 2
Completed | 3 | 2 | 1 | 2 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Left vLPFC cTBS/Right dlPFC iTBS/Left Som cTBS | Left vLPFC cTBS/Left Som cTBS/Right dlPFC iTBS | Left Som cTBS/Right dlPFC iTBS/Left vLPFC cTBS | Left Som cTBS/Left vLPFC cTBS/Right dlPFC iTBS | Right dlPFC iTBS/Left Som cTBS/Left vLPFC cTBS | Right dlPFC iTBS/Left vLPFC cTBS/Left Som cTBS | Total
Number analyzed (Participants) | 3 | 2 | 1 | 2 | 3 | 2 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 1 | 2 | 3 | 2 | 13
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 2 | 2 | 2 | 9
  Male | 2 | 0 | 1 | 0 | 1 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 2 | 2 | 1 | 2 | 2 | 2 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Brain Activity (Beta Power) in Left vLPFC
Description: The difference in brain activity (Beta power) in left vLPFC from pre TBS to post TBS. Higher numbers indicate more brain activity after TBS, while lower numbers indicate less brain activity (Beta power) after TBS.
Time Frame: Change in magnitude of brain activity (Beta power) immediately before and immediately after each TBS condition at EEG/TBS visits (15-30 mins)
Population: One participant was excluded from the EEG data analysis due to lack of immediate choices on the delayed discounting task
Measure: Mean (Standard Deviation); unit: Percentage of change post versus pre
Groups:
- Left vLPFC cTBS; Left SS cTBS: Continuous Theta Burst Stimulation (cTBS): cTBS is a brief stimulation of a part of the brain with a magnetic field that passes through the scalp and skull safely that can decrease the excitability of cortical neurons. It is FDA-approved as a treatment for psychological conditions including depression; however, this device is not approved for the treatment of adults with Bipolar Disorder I or for use in healthy adults. This research study is using the cTBS off label in all participants (those with and without Bipolar Disorder I) to examine research questions
- Right dlPFC iTBS: Intermittent Theta Burst Stimulation (iTBS): iTBS is a brief stimulation of a part of the brain with a magnetic field that passes through the scalp and skull safely to increase the excitability of cortical neurons. It is FDA-approved as a treatment for psychological conditions including depression; however, this device is not approved for the treatment of adults with Bipolar Disorder I or for use in healthy adults. This research study is using the cTBS off label in all participants (those with and without Bipolar Disorder I) to examine research questions.
Arm/Group | Left vLPFC cTBS | Right dlPFC iTBS | Left SS cTBS
Number analyzed (Participants) | 12 | 12 | 12
Percentage of change post versus pre
  Delayed Choice (larger reward in the future) | -88.78 (224.54) | 1437.64 (4411.75) | 13.43 (346.26)
  Immediate Choice (small immediate reward) | -128.00 (105.32) | -612.44 (1487.43) | 89.70 (940.52)
Statistical Analysis 1: Comparison: Left vLPFC cTBS; Paired t-test examining delayed choices on the delay discounting task (post versus pre). One participant was excluded from the EEG data analysis due to lack of immediate choices on the delay discounting task; Test type: Other; p = 0.29389090, t-test, 2 sided
Statistical Analysis 2: Comparison: Left vLPFC cTBS; Paired t-test examining immediate choices on the delay discounting task (post versus pre). One participant was excluded from the EEG data analysis due to lack of immediate choices on the delay discounting task; Test type: Other; p = 0.97863544, t-test, 2 sided
Statistical Analysis 3: Comparison: Right dlPFC iTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.60236264, t-test, 2 sided
Statistical Analysis 4: Comparison: Right dlPFC iTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.35845126, t-test, 2 sided
Statistical Analysis 5: Comparison: Left SS cTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.91766025, t-test, 2 sided
Statistical Analysis 6: Comparison: Left SS cTBS; Paired t-test examining immediate choices on the delayed discounting task (post versus pre). One participant was excluded from the EEG data analysis due to lack of immediate choices on the delayed discounting task; Test type: Other; p = 0.09605169, t-test, 2 sided

2. Primary Outcome: Brain Activity (Beta Power) in Right vLPFC
Description: The difference in brain activity (Beta power) in right vLPFC from pre TBS to post TBS. Higher numbers indicate more brain activity (Beta power) after TBS, while lower numbers indicate less brain activity (Beta power) after TBS.
Time Frame: as for outcome 1
Population: Initially, 10 main outcome measures were stated based on the assumption that 25 participants with bipolar disorder (BD) would be recruited and all data (neuroimaging and behavioral) would be collected from at least 20 participants. However, all data was collected from only 12 BD participants. As such, to not jeopardize the power for the 10 main outcome measures, statistical analyses were performed on only 4 of the 10 outcome measures.
Measure: Mean (Standard Deviation); unit: Percentage of change post versus pre
Arm/Group | Left vLPFC cTBS | Right dlPFC iTBS | Left SS cTBS
Number analyzed (Participants) | 12 | 12 | 12
Percentage of change post versus pre
  Delayed Choice (larger reward in the future) | -162.37 (799.00) | 5.13 (312.18) | -498.71 (1022.00)
  Immediate Choice (small immediate reward) | 131.99 (409.07) | -136.62 (702.68) | -117.6 (893.74)
Statistical Analysis 1: Comparison: Left vLPFC cTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.50030946, t-test, 2 sided
Statistical Analysis 2: Comparison: Left vLPFC cTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.37517380, t-test, 2 sided
Statistical Analysis 3: Comparison: Right dlPFC iTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.47876971, t-test, 2 sided
Statistical Analysis 4: Comparison: Right dlPFC iTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.21798816, t-test, 2 sided
Statistical Analysis 5: Comparison: Left SS cTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.47876971, t-test, 2 sided
Statistical Analysis 6: Comparison: Left SS cTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.21798816, t-test, 2 sided

3. Primary Outcome: Brain Activity (Beta Power) in Left dlPFC
Description: The difference in brain activity (Beta power) in left dLPFC from pre TBS to post TBS. Higher numbers indicate more brain activity (Beta power) after TBS, while lower numbers indicate less brain activity (Beta power) after TBS.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of change post versus pre
Arm/Group | Left vLPFC cTBS | Right dlPFC iTBS | Left SS cTBS
Number analyzed (Participants) | 12 | 12 | 12
Percentage of change post versus pre
  Delayed Choice (larger reward in the future) | 33.83 (446.73) | -286.13 (628.89) | -623.68 (1950.2)
  Immediate Choice (small immediate reward) | 32.04 (322.62) | -182.53 (494.97) | 99.64 (512.78)
Statistical Analysis 1: Comparison: Left vLPFC cTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.75298499, t-test, 2 sided
Statistical Analysis 2: Comparison: Left vLPFC cTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.16043787, t-test, 2 sided
Statistical Analysis 3: Comparison: Right dlPFC iTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.67902693, t-test, 2 sided
Statistical Analysis 4: Comparison: Right dlPFC iTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.33832977, t-test, 2 sided
Statistical Analysis 5: Comparison: Left SS cTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.67902693, t-test, 2 sided
Statistical Analysis 6: Comparison: Left SS cTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.33832977, t-test, 2 sided

4. Primary Outcome: Brain Activity (Beta Power) in Right dlPFC
Description: The difference in brain activity (Beta power) in right dLPFC from pre TBS to post TBS. Higher numbers indicate more brain activity (Beta power) after TBS, while lower numbers indicate less brain activity (Beta power) after TBS.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of change post versus pre
Arm/Group | Left vLPFC cTBS | Right dlPFC iTBS | Left SS cTBS
Number analyzed (Participants) | 12 | 12 | 12
Percentage of change post versus pre
  Immediate Choice (small immediate reward) | -128.27 (363.79) | -70.27 (520.40) | -383.76 (849.28)
  Delayed Choice (larger reward in the future) | -74.21 (104.49) | -83.74 (2072.87) | -398.00 (1039.5)
Statistical Analysis 1: Comparison: Left vLPFC cTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.73357221, t-test, 2 sided
Statistical Analysis 2: Comparison: Left vLPFC cTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.43954526, t-test, 2 sided
Statistical Analysis 3: Comparison: Right dlPFC iTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.44198980, t-test, 2 sided
Statistical Analysis 4: Comparison: Right dlPFC iTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.39565784, t-test, 2 sided
Statistical Analysis 5: Comparison: Left SS cTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.35602382, t-test, 2 sided
Statistical Analysis 6: Comparison: Left SS cTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.30499144, t-test, 2 sided

5. Primary Outcome: Functional Connectivity Between Left and Right vLPFC
Description: The difference in functional connectivity (a measure of interactions between 2 brain regions) among left and right vLPFC from preTBS to post TBS. Higher numbers indicate more functional connectivity after TBS, while lower numbers indicate less functional connectivity after TBS.
Time Frame: Change in magnitude of the functional connectivity immediately before and immediately after each TBS condition at EEG/TBS visits (15-30 mins)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of change post versus pre
Arm/Group | Left vLPFC cTBS | Right dlPFC iTBS | Left SS cTBS
Number analyzed (Participants) | 12 | 12 | 12
Percentage of change post versus pre
  Delayed Choice (larger reward in the future) | -0.34 (5.10) | -1.84 (4.92) | 0.36 (3.37)
  Immediate Choice (small immediate reward) | 3.26 (8.36) | -1.28 (6.19) | 1.07 (4.16)
Statistical Analysis 1: Comparison: Left vLPFC cTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.81601415, t-test, 2 sided
Statistical Analysis 2: Comparison: Left vLPFC cTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.20563452, t-test, 2 sided
Statistical Analysis 3: Comparison: Right dlPFC iTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.21947623, t-test, 2 sided
Statistical Analysis 4: Comparison: Right dlPFC iTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.45535329, t-test, 2 sided
Statistical Analysis 5: Comparison: Left SS cTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.21947623, t-test, 2 sided
Statistical Analysis 6: Comparison: Left SS cTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.45535329, t-test, 2 sided

6. Primary Outcome: Functional Connectivity Between vLPFC and Other RNet Regions
Description: The difference in functional connectivity (a measure of interactions between 2 brain regions) among vLPFC and other RNet regions from pre TBS to post TBS. Higher numbers indicate more functional connectivity after TBS, while lower numbers indicate less functional connectivity after TBS.
Time Frame: Change in magnitude of functional connectivity immediately before and immediately after each TBS condition at EEG/TBS visits (15-30 mins)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of change post versus pre
Arm/Group | Left vLPFC cTBS | Right dlPFC iTBS | Left SS cTBS
Number analyzed (Participants) | 12 | 12 | 12
Percentage of change post versus pre
  Delayed Choice (larger reward in the future) | 0.52 (6.68) | -1.03 (7.97) | -0.38 (4.99)
  Immediate Choice (small immediate reward) | 3.50 (8.29) | 0.69 (5.91) | 7.03 (7.58)
Statistical Analysis 1: Comparison: Left vLPFC cTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.83462055, t-test, 2 sided
Statistical Analysis 2: Comparison: Left vLPFC cTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.21582586, t-test, 2 sided
Statistical Analysis 3: Comparison: Right dlPFC iTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.59574875, t-test, 2 sided
Statistical Analysis 4: Comparison: Right dlPFC iTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.75948776, t-test, 2 sided
Statistical Analysis 5: Comparison: Left SS cTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.72384140, t-test, 2 sided
Statistical Analysis 6: Comparison: Left SS cTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.00477281, t-test, 2 sided

7. Primary Outcome: Functional Connectivity Between dlPFC With Other CEN Regions
Description: The difference in functional connectivity (a measure of interactions between 2 brain regions) among dlPFC and other RNet regions from pre TBS to post TBS. Higher numbers indicate more functional connectivity after TBS, while lower numbers indicate less functional connectivity after TBS.
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of change post versus pre
Arm/Group | Left vLPFC cTBS | Right dlPFC iTBS | Left SS cTBS
Number analyzed (Participants) | 12 | 12 | 12
Percentage of change post versus pre
  Delayed Choice (larger reward in the future) | 2.43 (5.64) | 2.03 (5.81) | 1.13 (6.16)
  Immediate Choice (small immediate reward) | -0.41 (4.47) | 3.86 (6.18) | 1.44 (6.17)
Statistical Analysis 1: Comparison: Left vLPFC cTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.20047055, t-test, 2 sided
Statistical Analysis 2: Comparison: Left vLPFC cTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.77922802, t-test, 2 sided
Statistical Analysis 3: Comparison: Right dlPFC iTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.29196708, t-test, 2 sided
Statistical Analysis 4: Comparison: Right dlPFC iTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.05605962, t-test, 2 sided
Statistical Analysis 5: Comparison: Left SS cTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.57368284, t-test, 2 sided
Statistical Analysis 6: Comparison: Left SS cTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.56397238, t-test, 2 sided

8. Secondary Outcome: Brain Activity (Beta Power) in Other RNet and CEN Regions
Description: The difference in brain activity (Beta power) among other RNet and CEN regions from pre TBS to post TBS. Higher numbers indicate more brain activity (Beta power) after TBS, while lower numbers indicate less brain activity (Beta power) after TBS.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of change post versus pre
Arm/Group | Left vLPFC cTBS | Right dlPFC iTBS | Left SS cTBS
Number analyzed (Participants) | 12 | 12 | 12
Percentage of change post versus pre
  Delayed Choice (larger reward in the future)(dorsal anterior cingulate cortex) | 248.65 (647.87) | -55.98 (124.11) | 41.73 (335.39)
  Immediate Choice (small immediate reward) (dorsal anterior cingulate cortex) | -45.54 (235.51) | -352.34 (1075.2) | 928.72 (2473.59)
  Delayed Choice (larger reward in the future) (posterior parietal cortex) | -77.80 (330.51) | 40.06 (217.51) | 142.64 (444.57)
  Immediate Choice (small immediate reward) (posterior parietal cortex) | -3.29 (65.09) | -89.97 (266.20) | -156.72 (289.48)
Statistical Analysis 1: Comparison: Left vLPFC cTBS; Paired t-test examining delayed choices on the delay discounting task (post versus pre) (dorsal anterior cingulate cortex). One participant was excluded from the EEG data analysis due to lack of immediate choices on the delay discounting task; Test type: Other; p = 0.86107891, t-test, 2 sided
Statistical Analysis 2: Comparison: Left vLPFC cTBS; Paired t-test examining immediate choices on the delay discounting task (post versus pre) (dorsal anterior cingulate cortex). One participant was excluded from the EEG data analysis due to lack of immediate choices on the delay discounting task; Test type: Other; p = 0.62228799, t-test, 2 sided
Statistical Analysis 3: Comparison: Right dlPFC iTBS; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.79477883, t-test, 2 sided
Statistical Analysis 4: Comparison: Right dlPFC iTBS; [analysis description as in outcome 8, analysis 2]; Test type: Other; p = 0.12634435, t-test, 2 sided
Statistical Analysis 5: Comparison: Left SS cTBS; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.79477883, t-test, 2 sided
Statistical Analysis 6: Comparison: Left SS cTBS; [analysis description as in outcome 8, analysis 2]; Test type: Other; p = 0.12634435, t-test, 2 sided
Statistical Analysis 7: Comparison: Left vLPFC cTBS; Paired t-test examining delayed choices on the delay discounting task (post versus pre) (posterior parietal cortex). One participant was excluded from the EEG data analysis due to lack of immediate choices on the delay discounting task; Test type: Other; p = 0.62461968, t-test, 2 sided
Statistical Analysis 8: Comparison: Left vLPFC cTBS; Paired t-test examining immediate choices on the delay discounting task (post versus pre) (posterior parietal cortex). One participant was excluded from the EEG data analysis due to lack of immediate choices on the delay discounting task; Test type: Other; p = 0.51324793, t-test, 2 sided
Statistical Analysis 9: Comparison: Right dlPFC iTBS; [analysis description as in outcome 8, analysis 7]; Test type: Other; p = 0.60543603, t-test, 2 sided
Statistical Analysis 10: Comparison: Right dlPFC iTBS; [analysis description as in outcome 8, analysis 8]; Test type: Other; p = 0.75565448, t-test, 2 sided
Statistical Analysis 11: Comparison: Left SS cTBS; [analysis description as in outcome 8, analysis 7]; Test type: Other; p = 0.60543603, t-test, 2 sided
Statistical Analysis 12: Comparison: Left SS cTBS; [analysis description as in outcome 8, analysis 8]; Test type: Other; p = 0.75565448, t-test, 2 sided

9. Secondary Outcome: Functional Connectivity Among Other RNet and CEN Regions
Description: The difference in functional connectivity (a measure of interactions between 2 brain regions) among other RNet and CEN regions from pre TBS to post TBS. Higher numbers indicate more functional connectivity after TBS, while lower numbers indicate less functional connectivity after TBS.
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of change post versus pre
Arm/Group | Left vLPFC cTBS | Right dlPFC iTBS | Left SS cTBS
Number analyzed (Participants) | 12 | 12 | 12
Percentage of change post versus pre
  Delayed Choice (larger reward in the future)(Left vLPFC and Posterior Parietal Cortex) | 2.45 (4.33) | -2.10 (7.23) | 1.18 (4.97)
  Immediate Choice (small immediate reward) (Left vLPFC and Posterior Parietal Cortex) | 2.33 (9.95) | 3.83 (13.52) | 1.27 (7.24)
Statistical Analysis 1: Comparison: Left vLPFC cTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.09266386, t-test, 2 sided
Statistical Analysis 2: Comparison: Left vLPFC cTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.53980185, t-test, 2 sided
Statistical Analysis 3: Comparison: Right dlPFC iTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.30223686, t-test, 2 sided
Statistical Analysis 4: Comparison: Right dlPFC iTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.39166649, t-test, 2 sided
Statistical Analysis 5: Comparison: Left SS cTBS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.30223686, t-test, 2 sided
Statistical Analysis 6: Comparison: Left SS cTBS; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.39166649, t-test, 2 sided

10. Secondary Outcome: Immediate Choices Made on the Delay Discounting Task
Description: The sum (overall total) of the immediate choices (choosing to receive a small immediate reward) made on the delay discounting task
Time Frame: 15-30 minutes
Measure: Mean (Standard Deviation); unit: percentage of immediate choices changes
Arm/Group | Left vLPFC cTBS | Right dlPFC iTBS | Left SS cTBS
Number analyzed (Participants) | 13 | 13 | 13
percentage of immediate choices changes | -18.47 (29.74) | -9.78 (29.74) | -26.28 (27.38)
Statistical Analysis 1: Comparison: Left vLPFC cTBS; Paired t-test (post versus pre); Test type: Other; p = 0.0265, t-test, 2 sided
Statistical Analysis 2: Comparison: Right dlPFC iTBS; Paired t-test (post versus pre); Test type: Other; p = 0.1053, t-test, 2 sided
Statistical Analysis 3: Comparison: Left SS cTBS; Paired t-test (post versus pre); Test type: Other; p = 0.0033, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Total participation up to 1 day
Groups:
- Left Som cTBS: Continuous Theta Burst Stimulation (cTBS): cTBS is a brief stimulation of a part of the brain with a magnetic field that passes through the scalp and skull safely that can decrease the excitability of cortical neurons. It is FDA-approved as a treatment for psychological conditions including depression; however, this device is not approved for the treatment of adults with Bipolar Disorder I or for use in healthy adults. This research study is using the cTBS off label in all participants (those with and without Bipolar Disorder I) to examine research questions
Arm/Group | Left vLPFC cTBS | Right dlPFC iTBS | Left Som cTBS
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT05179785/Prot_SAP_002.pdf